CLINICAL TRIAL: NCT00255723
Title: Risk-Adapted High Dose Chemoradiotherapy and Autologous Stem Cell Transplantation for Patients With Relapsed and Primary Refractory Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients Who Are Undergoing an Autologous Stem Cell Transplant for Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-047; MSKCC-04047
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma
Keywords: adult lymphocyte depletion Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Carboplatin; Etoposide; Ifosfamide

ARMS (2):
- Cytoreductive chemotherapy group 1 (Experimental): Patients receive ICE comprising ifosfamide IV and carboplatin IV once on day 2 and etoposide IV over 1 hour once daily on days 1-3. Patients then receive ifosfamide IV twice on day 15, carboplatin IV once on day 17 and etoposide IV over 1 hour twice daily on days 15-17.
  Interventions: Drug: carboplatin; Drug: etoposide; Drug: ifosfamide
- Cytoreductive chemotherapy group 2 (Experimental): Patients receive ifosfamide IV twice on days 1 and 17, carboplatin IV once on days 3 and 19, and etoposide IV over 1 hour twice daily on days 1-3 and 17-19.
  Interventions: Drug: carboplatin; Drug: etoposide; Drug: ifosfamide

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: etoposide — Given IV
Drug: ifosfamide — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Radiation therapy uses high-energy x-rays to kill cancer cells. Giving combination chemotherapy and radiation therapy with an autologous stem cell transplant, using peripheral stem cells or bone marrow from the patient, may allow more chemotherapy to be given so that more cancer cells are killed. Giving combination chemotherapy together with radiation therapy before an autologous stem cell transplant may be an effective treatment for Hodgkin's lymphoma.

PURPOSE: This phase II trial is studying how well combination chemotherapy and radiation therapy work in treating patients who are undergoing an autologous stem cell transplant for relapsed or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether event-free survival of patients with low to high-intermediate risk, relapsed or refractory Hodgkin's lymphoma can be improved when treated with cytoreductive combination chemotherapy followed by radiotherapy, high-dose combination chemotherapy, and autologous stem cell transplantation.

Secondary

* Determine the toxic effects of this regimen in these patients.

OUTLINE: Patients are stratified according to risk factors (low or low-intermediate risk [0-1 risk factor] vs high-intermediate risk [2 risk factors]).

* ICE-based cytoreductive chemotherapy: Patients are assigned to 1 of 2 treatment groups.

  * Group I (patients with low or low-intermediate risk disease): Patients receive ICE comprising ifosfamide IV and carboplatin IV once on day 2 and etoposide IV over 1 hour once daily on days 1-3. Patients then receive ifosfamide IV twice on day 15, carboplatin IV once on day 17 and etoposide IV over 1 hour twice daily on days 15-17.
  * Group II (patients with high-intermediate risk disease): Patients receive ifosfamide IV twice on days 1 and 17, carboplatin IV once on days 3 and 19, and etoposide IV over 1 hour twice daily on days 1-3 and 17-19.

In both groups, patients undergo stem cell collection after either the first or second OR first and second courses of ICE.

* Stem cell mobilization and collection: Patients receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 5 and continuing until stem cell collection is completed. Patients undergo a maximum of 5 daily apheresis sessions. Patients who mobilize fewer than the required minimal number of stem cells repeat apheresis with high-dose G-CSF alone or undergo bone marrow harvest. Patients then proceed to radiotherapy, high-dose chemotherapy (HDC), and autologous stem cell transplant (ASCT) OR noncross-resistant chemotherapy based on response to ICE-based cytoreductive chemotherapy.
* Restaging studies: Patients undergo restaging studies with CT scan and positron emission tomography (PET). Patients who are chemosensitive with a normal PET scan proceed to radiotherapy, HDC, and ASCT. Patients who progress on ICE, or who respond but have an abnormal PET scan, proceed to noncross-resistant chemotherapy comprising gemcitabine hydrochloride, vinorelbine, and doxorubicin HCl liposome (GND).
* GND chemotherapy: Patients receive gemcitabine hydrochloride IV, vinorelbine IV, and doxorubicin HCl liposome IV on days 1, 15, 29, and 43. Patients then proceed to radiotherapy, HDC, and ASCT in the absence of disease progression.
* Radiotherapy: Within 2 weeks after completion of the ICE or GND regimen, patients who have no history of prior radiotherapy receive radiotherapy according to stratification by disease extent (isolated lymph nodes vs ≥ 2 contiguous nodal-based masses with or without extensive small-volume lymphadenopathy vs extensive small-volume lymphadenopathy). These patients undergo either involved-field radiotherapy (IFRT) twice daily over 1-2 weeks, total lymphoid irradiation (TLI) twice daily over 1 week, or both concurrently.
* HDCT: Patients who undergo TLI only OR IFRT and TLI receive high-dose cyclophosphamide IV twice daily and etoposide IV once daily on days -5 and -2. Patients who undergo IFRT only OR do not undergo radiotherapy receive high-dose cyclophosphamide IV twice daily and etoposide IV once daily on days -6 and -3 and carmustine IV once on day -2.
* ASCT: Patients undergo ASCT or reinfusion of bone marrow, if harvested, on day -1 or 0. Patients then receive G-CSF beginning on day 5 and continuing until blood counts recover.

After completion of study treatment, patients are followed periodically for 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of Classical Hodgkin's Lymphoma. Lymphocyte predominant histology will be excluded.
* Primary refractory or relapsed disease proven by biopsy or fine needle aspiration (cytology) of an involved site
* Failure of doxorubicin or nitrogen mustard containing front-line therapy
* 18F-fluorodeoxyglucose-PET scan demonstrating PET avid disease
* Cardiac ejection fraction of greater than 45%, measured since last chemotherapy.
* Adjusted diffusing capacity of greater than 50% on pulmonary function testing, measured since last chemotherapy
* Serum creatinine < than or = to 1.5 mg/dl; if creatinine >1.5 mg/dl then the measured 12- or 24-hour creatinine clearance must be >60 ml/minute.
* ANC>1000/μl and Platelets>50,000/μl
* Total bilirubin < than or = to 2.0 mg/dl in the absence of a history of Gilbert's disease.
* Females of childbearing age must be on an acceptable form of birth control.
* Age between 18 and 72
* HIV I and II negative.
* Patients or their guardians must be capable of providing informed consent.

Exclusion Criteria:

Histology for Lymphocyte predominant subtype Hodgkin's Lymphoma

* Prior treatment with carboplatin, cisplatin, ifosfamide, gemcitabine, or vinorelbine
* Hepatitis B surface antigen positive.
* Known pregnancy or breast-feeding.
* Medical illness unrelated to Hodgkin's Lymphoma, which, in the opinion of the attending physician and/or principal investigator, will preclude administering chemotherapy safely.
* History of any malignancy for which the disease-free interval is <5 years, excluding curatively treated cutaneous basal cell or squamous cell carcinoma and carcinoma in-situ of the cervix

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Moskowitz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Driessen J, Zwezerijnen GJC, Schoder H, Kersten MJ, Moskowitz AJ, Moskowitz CH, Eertink JJ, Heymans MW, Boellaard R, Zijlstra JM. Prognostic model using 18F-FDG PET radiomics predicts progression-free survival in relapsed/refractory Hodgkin lymphoma. Blood Adv. 2023 Nov 14;7(21):6732-6743. doi: 10.1182/bloodadvances.2023010404. PMID 37722357
- [Derived] Moskowitz CH, Matasar MJ, Zelenetz AD, Nimer SD, Gerecitano J, Hamlin P, Horwitz S, Moskowitz AJ, Noy A, Palomba L, Perales MA, Portlock C, Straus D, Maragulia JC, Schoder H, Yahalom J. Normalization of pre-ASCT, FDG-PET imaging with second-line, non-cross-resistant, chemotherapy programs improves event-free survival in patients with Hodgkin lymphoma. Blood. 2012 Feb 16;119(7):1665-70. doi: 10.1182/blood-2011-10-388058. Epub 2011 Dec 19. PMID 22184409

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Standard dose ICE x 1 cycle, followed by augmented ICE x 1 cycle (0-1 risk factors)
- Arm B: Augmented ICE x 2 cycles (2 risk factors)
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 56 | 41
Completed | 54 | 39
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1
Not completed — Response Data Not Available | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 56 | 41 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 55 | 38 | 93
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 21 | 56
  Male | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Overall objective response to therapy Complete remission/unconfirmed (CRu)
  This includes patients who meet criteria for CR with the following exceptions:
  1. A residual lymph node mass > 1.5 cm in the short axis with normalization of 18Ffluorodeoxyglucose- PET scan Partial remission/minimal response (PR and MR)
  1. Any decrease in lymph nodes and nodal-based masses
  2. Any decrease in PET avidity (however, residual FDG uptake is present)
  3. Involving organs involved prior to therapy must have diminished in size.
  4. No new sites of disease Stable disease Response is less than that which constitutes a PR and disease does not meet criteria for progressive disease Progressive disease
  1. Increase in lymph nodes or nodal-based masses, or other measurable disease from pretreatment observations. 2. Appearance of any new lesion at the end of therapy
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 54 | 39
participants
  Complete Remission | 45 | 31
  Partial Remission (PR) | 6 | 1
  Progression of Disease (POD) | 3 | 7

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 8/56 | 18/41
Other Adverse Events (participants affected / at risk) | 56/56 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=56) | Arm B (N=41)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome/acute infusion reaction (General disorders) | 1 (1) | 0 (0)
Death not associated with CTCAE term- Death NOS (General disorders) | 0 (0) | 1 (1)
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Febrile neutropenia (General disorders) | 1 (2) | 4 (4)
Catheter related infection (Infections and infestations) | 2 (2) | 4 (4)
Infective myositis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (2) | 0 (0)
Infection, other (Infections and infestations) | 1 (1) | 0 (0)
Large intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain - Chest/thorax NOS (General disorders) | 1 (1) | 0 (0)
Pericardial effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vascular- Other (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=56) | Arm B (N=41)
ALT, SGPT (Blood and lymphatic system disorders) | 7 (7) | 4 (4)
AST, SGOT (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 10 (10) | 10 (10)
Hemoglobin (Blood and lymphatic system disorders) | 49 (49) | 39 (39)
Prothrombin Time and International Normalized Ratio (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 55 (55) | 39 (39)
Lymphopenia (Blood and lymphatic system disorders) | 55 (55) | 41 (41)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 55 (55) | 39 (39)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 38 (38) | 23 (23)
Platelets (Blood and lymphatic system disorders) | 55 (55) | 38 (38)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 24 (24) | 17 (17)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 16 (16) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes